CLINICAL TRIAL: NCT00728793
Title: A Phase I Open-Label, Multiple Dose, Sequential Dose Escalation Study to Investigate the Safety and Pharmacokinetics of Intravenous CUDC-101 in Subjects With Advanced and Refractory Solid Tumors
Brief Title: A Phase I Study of the Safety, Pharmacokinetics, and Anti-Tumor Activity of CUDC-101 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-101-101
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2015-09

CONDITIONS: Tumors
Keywords: Advanced Solid Tumors; EGFR; HDAC; Her2; Open-Label; Dose-Escalation
MeSH Terms: conditions — Neoplasms | interventions — 7-(4-(3-ethynylphenylamino)-7-methoxyquinazolin-6-yloxy)-N-hydroxyheptanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CUDC-101 — Doses will be given by intravenous infusion over 1 hour on days 1-5 of each treatment cycle. Total treatment cycle duration will be 14 days. Additional treatment cycles will be administered until the subjects withdraws consent, experiences unacceptable toxicity, or if there is documented tumor progression.

SUMMARY:
This is a phase I, open-label, dose-escalation study of CUDC-101 in patients with advanced and refractory solid tumors. CUDC-101 is a multi-targeted agent designed to inhibit epidermal growth factor receptor (EGFR), human epidermal growth factor receptor Type 2(Her2) and histone deacetylase (HDAC). The study is designed to establish the safety, including the maximum tolerated dose, the pharmacokinetics, and the anti-tumor activity of CUDC-101.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced, refractory solid tumors and a histopathologically confirmed diagnosis
* Subjects must have no further standard of care options or have refused standard therapy
* Measurable or evaluable disease
* Age ≥ 18 years
* ECOG performance < 2
* Life expectancy ≥ 3 months
* If female, neither pregnant or lactating
* If of child bearing potential, must use adequate birth control
* Absolute neutrophil count ≥ 1,500/µL; platelets ≥ 100,000/µL;
* Creatinine ≤ 1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60mL/min/1.73m2
* Total bilirubin ≤ 1.5x ULN; AST/ALT ≤ 2.5x ULN. In subjects with documented liver metastases, the AST/ALT may be ≤ 5x ULN
* Prothrombin time ≤1.5x ULN, unless receiving therapeutic anticoagulation
* Serum magnesium and potassium within normal limits (may be supplement to achieve normal values)
* Subjects with brain metastases are eligible if controlled on a stable dose ≤ 10mg prednisone/day or its equivalent dose of steroids
* Able to render informed consent and to follow protocol requirements.

Exclusion Criteria:

* Anticancer therapy within 4 weeks of study entry. Prostate cancer subjects on LHRH hormonal therapy may be enrolled and continue on this therapy.
* Use of investigational agent(s) within 30 days of study entry
* History of cardiac disease with a New York Heart Association (NYHA) Class II or greater congestive heart failure (CHF), myocardial infarction (MI) or unstable angina in the past 6 months prior to Day 1 of treatment, serious arrhythmias requiring medication for treatment.
* Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
* The following are permitted but should be used with caution and other suitable agents used if possible:

  * Subjects receiving concomitant medications metabolized by CYP 3A4 and CYP 2D6
  * CYP3A4 inducers
  * CYP3A4 inhibitors
  * Warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The highest dose level of CUDC-101 at which <33% of at least 6 or more subjects experiences a dose limiting toxicity. | Study treatment period - approximately 12 months
  The maximum tolerated dose is the highest dose level at which <33% of at least 6 or more subjects experiences a dose limiting toxicity.
The number of patients with adverse events. | Study treatment period - approximately 12 months
  The number of patients with adverse events will be assessed to determine the safety and tolerability of CUDC-101.

SECONDARY OUTCOMES:
Number of patients that show a response (complete response or partial response) based on RECIST criteria. | Study treatment period - approximately 12 months
  To evaluate the efficacy of CUDC-101 in subjects with advanced and refractory solid tumors, responses based on RECIST criteria will be evaluated.
Plasma concentration of CUDC-101 over time from Day 1 through Day 6. | Approximately 1 week
  To assess the pharmacokinetics of CUDC-101 in this patient population, plasma concentration of CUDC-101 will be measured over time from Day 1 through Day 6.
Measurement of epidermal growth factor receptor (EGFR) in archival tumor tissue, skin biopsies and tumor biopsies. | Pre-treatment through Day 5 of cycle 1 - approximately 1 week
  Measurement of EGFR to evaluate pharmacodynamic biomarkers of CUDC-101 activity.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tolcher, M.D., Principal Investigator — START (South Texas Accelerated Research Therapeutics)
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - START (South Texas Accelerated Research Therapeutics), San Antonio, Texas

REFERENCES:
- See also: Curis, Inc. Company Website — http://www.curis.com